CLINICAL TRIAL: NCT05460104
Title: Impact of the Use of Virtual Reality Exposure Therapy on Body Image After Bariatric Surgery
Brief Title: Impact of the Use of VERT on Body Image After Bariatric Surgery
Acronym: BARIAREV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2021/37
Record Dates: First submitted 2022-06-15; First posted 2022-07-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: Virtual Reality Exposure Therapy; Body image; Dysmorphophobia
MeSH Terms: conditions — Obesity; Body Dysmorphic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expérimental (Experimental): Virtual Reality Exposure Therapy will be realised.
  Interventions: Device: Experimental
- Control (Active Comparator): Standard care without VRET
  Interventions: Other: Control

INTERVENTIONS:
Device: Experimental — Virtual reality sessions with a psychologist (30 minutes per session) once a week for 10 weeks. Work of the psychologist on a virtual environment created for the protocol in partnership with the company.
  Arms: Expérimental
Other: Control — Standard care is medical follow-up, no specific psychological care.
  Arms: Control

SUMMARY:
The purpose ot the study is to assess the effectiveness of the use of VERT on improving body image at 12 months in patients who underwent bariatric surgery in the weight stabilization phase (between 18 and 30 months after bariatric) presenting dissatisfaction with their body image compared to standard follow-up in post-bariatric surgery (lack of specific management of body image).

DETAILED DESCRIPTION:
Virtual reality therapy makes it possible to work on the integration of proprioceptive information via the reproduction of environments close to reality and therefore allow the patient to accept his new identity. This tool is used in an increasing number of indications and in particular in the management of dysmorphophobia in patients suffering from anorexia nervosa. In the context of bariatric surgery, only case reports have been published so far. Significant improvements in the body satisfaction scores of patients have been showed, in patients who had undergone bariatric surgery who presented bodily dissatisfaction after 6 weeks of virtual reality. However, larger numbers, longer follow-up periods and more rigorous methodologies are needed to confirm the impact of this practice. The hypothesis of the study is that virtual reality therapy could improve body image in patients who are dissatisfied with their body image after bariatric surgery.

ELIGIBILITY:
* inclusion criteria: patients who underwent bariatric surgery in the weight stabilization phase (between 18 and 30 months after surgery) presenting dissatisfaction with their body image according to the BSQ (score ≥ 111), to be affiliated to the French social security system. The prior, free and informed consent of the patient shall be obtained.
* exclusion criteria: patients with disabling nausea (Motion Sickness) from previous use of a virtual reality headset, patients who had from post-bariatric reconstructive surgery, epileptic patients, decompensation of a psychiatric pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-12-19 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Body Shape Questionnaire | Between inclusion and 12 months after.
  Average variation of the Body Shape Questionnaire (BSQ). BSQ is a 34 questions questionnaire, for each question the answer is 1 to 6, 1 for "never" and 6 for "always".
  (score ≥ 111, moderate body image concern)

SECONDARY OUTCOMES:
Change weight | Between inclusion day and Month 3
  Average weight loss in %, in the two arms.
Change weight | Between Month 6 and Month 12
  Average weight loss in %, in the two arms.
Body Image Assessment for Obesity questionnaire | Between inclusion day and Month 3
  Average variation in Body Image Assessment for Obesity, in each arm. The patient surrounds the figure that seems to closest to his or her current figure. And then he surrounds the figure he would like to achieve.This is a schematic representation of the body, from the thinnest silhouette in 1 to the widest in 18
Body Image Assessment for Obesity questionnaire | Between Month 6 and Month 12
  Average variation in Body Image Assessment for Obesity questionnaire, in each arm.The patient surrounds the figure that seems to closest to his or her current figure. And then he surrounds the figure he would like to achieve. This is a schematic representation of the body, from the thinnest silhouette in 1 to the widest in 18
Quality of Life, Obesity and Dietetics questionnaire assess quality of life | Between inclusion day and Month 3
  Average variation of the Quality of Life, Obesity and Dietetics, in each arm. This questionnaire consists of 36 questions that focus on the effects of the weight problem as experienced by the patient. For each question the patient can answer from 1 to 5: 1 always, 5 never.
Quality of Life, Obesity and Dietetics questionnaire assess quality of life | Between Month 6 and Month 12
  Average variation of the Quality of Life, Obesity and Dietetics, in each arm. This questionnaire consists of 36 questions that focus on the effects of the weight problem as experienced by the patient. For each question the patient can answer from 1 to 5: 1 always, 5 never.
Self-esteem | Between inclusion day and Month 3
  Average variation of the Rosenberg Self-Esteem Scale, in each arm. The scale represents an assessment of the person's overall self-esteem. The scale consists of 10 statements measured on a scale of 1 to 4: 1 "Totally disagree", 4 "Totally agree".
  The score is between 10 and 40. A score below 25 indicates very low self-esteem. A score between 25 and 31 indicates low self-esteem. A score between 31 and 34 indicates average self-esteem. A score between 34 and 39 indicates strong self-esteem. A score above 39 indicates very high self-esteem.
Self-esteem | Between Month 6 and Month 12
  Average variation of the Rosenberg Self-Esteem Scale, in each arm.The scale represents an assessment of the person's overall self-esteem. The scale consists of 10 statements measured on a scale of 1 to 4: 1 "Totally disagree", 4 "Totally agree".
  The score is between 10 and 40. A score below 25 indicates very low self-esteem. A score between 25 and 31 indicates low self-esteem. A score between 31 and 34 indicates average self-esteem. A score between 34 and 39 indicates strong self-esteem. A score above 39 indicates very high self-esteem.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CH de Libourne - Hôpital Robert BOULIN, Libourne
  - CHU de Bordeaux - Hopital Haut-Lévêque, Pessac

IPD SHARING:
Plan to Share IPD: No